CLINICAL TRIAL: NCT00855283
Title: Intranasal Administration of Neostigmine and Glycopyrrolate for Bowel Evacuation
Brief Title: Intranasal Administration of a Prokinetic for Bowel Evacuation in Persons With SCI
Acronym: IN NEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4162C-2; KOR-11-018 (Other: James J. Peters VA Medical Center)
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: SCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): SCI
  Interventions: Drug: IN NEO; Drug: IN NEO + IN Glycopyrrolate; Drug: IV Visit

INTERVENTIONS:
Drug: IN NEO — 20 mg Neostigmine via intranasal and sublingual administration
Drug: IN NEO — 40 mg Neostigmine via intranasal administration
Drug: IN NEO — 60 mg Neostigmine via intranasal administration
Drug: IN NEO + IN Glycopyrrolate — Intranasal or sublingual Neostigmine (at effective dose: 20, 40, or 60 mg) + 4-12 mg intranasal or sublingual Glycopyyrolate
Drug: IV Visit — 2mg NEO and .4mg GLY given intravenously to see if the subject responds to the intervention. If they respond, then they will proceed to the IN portion of the study.

SUMMARY:
DWE (difficulty with evacuation) is a common and an important quality of life issue after spinal cord injury. Not only is the management DWE time-consuming and unpleasant, but the results are often suboptimal in terms of complications such as incontinence and impaction. Bowel care regimens after spinal cord injury have not changed in any significant fashion in many years. The usual strategies for attaining bowel evacuation involve dietary manipulation (e.g., high fiber diets and hydration), thrice weekly laxative administration (senna and cascara) and thrice weekly anorectal instillation of cathartics (enemas and suppositories). Bowel care can be quite time consuming (greater than 2 hours in many instances) and may also require extensive nursing care. Finally, incomplete evacuation could contribute to fecal incontinence that has significant morbidity in these patients.

In preliminary studies performed at the JJPVAMC, IV, IM, and subcutaneous injection of neostigmine combined with glycopyrrolate were demonstrated to be highly effective to promote bowel evacuation in the SCI population. In an effort to provide a more realistic administration of this procedure, we propose to test the intranasal spray injection of neostigmine and glycopyrrolate for safety and efficacy.

DETAILED DESCRIPTION:
We have been studying the effects of spinal cord injury on the bowel for over ten years. Our data suggests that one of the fundamental consequences of spinal cord injury is a slowing of intestinal peristaltic activity, most likely as a result of down regulation of parasympathetic neural pathways. Furthermore, measures that increase parasympathetic stimulation to the bowel result in bowel evacuation and improve bowel care. In this respect, significant acute effects have been demonstrated after the intravenous administration of the cholinergic agent neostigmine (Am J Gastro 100:1560-5, 2005). Long term efficacy has also been shown using intramuscular administration of neostigmine (Gastro 128:P258, 2005). Subcutaneous administration of neostigmine is in progress at this time. Bowel evacuation also is facilitated by subcutaneous administration but often requires a second dose (30 minutes after the first). This observation is likely due to a decreased rate of absorption from this tissue compartment and a correspondingly lower peak level of neostigmine (vide infra). Given the potential cardiopulmonary toxicity of neostigmine (bradycardia and bronchoconstriction), neostigmine was administered in these studies in combination with the anticholinergic agent glycopyrrolate. We have reported that the latter selectively blocks the cardiopulmonary side effects of neostigmine without significantly decreasing the prokinetic peristaltic response. In summary, our data to date indicates that the combined administration of neostigmine and glycopyrrolate is safe after spinal cord damage and it results in predicable and prompt bowel evacuation.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete or complete SCI
* Tetraplegia or paraplegia
* Males or females
* Age 18 (no upper age limit)
* Excess time for bowel evacuation (> 60 minutes per bowel training session)

Exclusion Criteria:

* Persons with SCI who do not require do not require additional bowel care or have "normal bowel function"
* Known hypersensitivity to neostigmine or glycopyrrolate
* History of mechanical obstruction of the intestine or urinary tract.
* Myocardial infarction within less than 6 months of trial.
* Hemodynamic instability
* Potential for pregnancy. (Women who are sexually active and of childbearing potential (i.e. not surgically sterile or at least 2 year postmenopausal) must be have a negative serum pregnancy test and to have utilized one of the following methods of contraception prior to screening: barrier (condom, diaphragm with spermicide) intrauterine device, or tubal ligation beginning at least 30 days prior; hormonal (oral, injectable, transdermal, or implanted) beginning at least 3 months prior; or vasectomized partner for at least the prior 6 months. Subjects must agree to maintain these contraceptive methods through the completion of the study.)
* Lactating/nursing females
* Patients who develop significant bradycardia (HR<42 bpm) or other significant anticholinergic symptoms (e.g., severe cramps, dry mouth, etc.) any time during the study will be discontinued.
* Concurrent participation in other clinical trials (within 30 days).
* Use of concurrent medications that affect cardiac output (e.g. tricyclics, beta blockers, etc.)
* Fluctuating use of concurrent medications (should be stable for 3-4 weeks before and no changes anticipated throughout the study).
* History of reduced cardiac output (via history and ECG) in addition to myocardial infarction and hemodynamic instability.
* Concurrent history of peripheral vascular disease, kidney disease, etc.
* Asthma or other broncho-constrictive disorders.
* Hemoglobin level < 12 g/dL

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bowel evacuation | <60 min

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Korsten, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States